CLINICAL TRIAL: NCT06174623
Title: Early Feasibility Study to Mechanically Support Cardiorenal Function in Acute Decompensated Heart Failure With Diuretic Resistance
Brief Title: Feasibility Study to Support Cardiorenal Function in Acute Decompensated Heart Failure With Diuretic Resistance
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Puzzle Medical Devices Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MH-ADHF-001
Record Dates: First submitted 2023-11-30; First posted 2023-12-18 (Actual); Last update posted 2024-06-17 (Actual); Status verified 2024-06

CONDITIONS: Heart Failure; Acute Decompensated Heart Failure; Cardiorenal Syndrome; Heart Failure, Congestive; Heart Failure With Preserved Ejection Fraction; Heart Failure With Reduced Ejection Fraction; Diuretic Resistance
Keywords: Puzzle Medical Devices; ModulHeart; Mechanical Circulatory Support; Intra-Aortic; MCS; LVAD; pVAD; percutaneous ventricular assist device; Left ventricular assist device
MeSH Terms: conditions — Heart Failure; Cardio-Renal Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ModulHeart System (Experimental)
  Interventions: Device: ModulHeart Support

INTERVENTIONS:
Device: ModulHeart Support — The ModulHeart device will be implanted in the descending abdominal aorta.

SUMMARY:
Evaluation of the safety and efficacy of the ModulHeart System in patients hospitalized with acute decompensated heart failure (ADHF) and diuretic resistance

DETAILED DESCRIPTION:
The study is a prospective, single-arm, non-randomized feasibility study to evaluate the safety and performance of the ModulHeart System in patients hospitalized with ADHF and diuretic resistance. The ModulHeart system consists of the ModulHeart Delivery System, the ModulHeart Pumps, the ModulHeart Controller, and the ModulHeart Retrieval System.

ELIGIBILITY:
Inclusion Criteria:

1. Admitted to the hospital with a primary diagnosis of ADHF
2. Clinical signs and/or symptoms of congestion defined as at least one of the following: dyspnea at rest or with minimal exertion, orthopnea, lower extremity edema (≥2+), elevated jugular venous pressure, pulmonary rales, pulmonary vascular congestion on chest x-ray, pleural effusion or ascites
3. Projected need by the treating clinician for continued treatment with IV diuretic agents for more than 48 hours with the goal of significant fluid removal (more than 1L net fluid loss/24h)
4. Appropriate intravenous loop diuretic therapy at the time of enrollment, defined as at least the higher of:

   1. Furosemide 40mg IV bid or equivalent
   2. IV furosemide or equivalent IV loop diuretic equivalent to ≥2x the total oral daily loop diuretic dose at home in 2 divided doses
5. Diuretic resistance defined as at least ONE of the following:

   1. Urine output of less than 1.5L over 12h following the last diuretic dose, OR
   2. Net fluid loss of less than 1L over the last 24 hours, OR
   3. Spot urinary sodium concentration of less than 70 mmol/L 2h following the last diuretic dose or cumulative 6-hour natriuresis of less than 100 mmol following the last diuretic dose, OR
   4. Clinically unsatisfactory resolution of congestion
6. Age ≥ 21 years old
7. Signed informed consent

Exclusion Criteria:

1. ADHF related to acute secondary disease (i.e., infection or acute coronary syndrome)
2. Treatment with high dose inotropes (milrinone ≥0.375 mcg/kg/min, dobutamine ≥5mcg/kg/min or dopamine ≥5mcg/kg/min) and/or treatment with vasopressors to maintain a systolic arterial blood pressure ≥90 mmHg or mean arterial blood pressure ≥60 mmHg
3. Current or previous support with a durable left ventricular assist device (LVAD) at any time or use of an extracorporeal membrane oxygenation (ECMO), percutaneous ventricular assist devices, intra-aortic balloon pump or patient on home inotropes currently or within the last 30 days
4. Recent myocardial infarction, percutaneous coronary intervention or surgical revascularization (within the last 30 days) or awaiting planned coronary intervention or surgery
5. Fixed pulmonary vascular resistance of more than 5 Wood units, estimated PASP of more than 80 mmHg as measured on echocardiogram or echocardiographic evidence of primarily right heart failure
6. Prior heart transplant, heart failure due to rejection of a previous heart transplant, or planned heart transplantation
7. Reanimated cardiac arrest in the last 30 days
8. Suspected or known amyloid disease or other restrictive cardiomyopathy
9. Severe bleeding risk precluding anticoagulation:

   1. Previous intracranial bleed unless there is documentation in the medical record (from a physician that is not part of the study) that the patient can safely use anticoagulation for 3 days
   2. Gastrointestinal (GI) bleeding within 1 month requiring hospitalization and/or transfusion
   3. Recent major surgery within 1 month if the surgical wound is judged to be associated with an increased risk of bleeding
   4. Platelet count of less than 50,000 cells/mm3
   5. Uncorrectable bleeding diathesis or coagulopathy
10. Contraindicated anatomy:

    1. Descending aortic anatomy that would prevent safe placement of the device (less than 18 mm or more than 28mm thoracoabdominal aorta diameter at deployment location)
    2. Abnormalities of the aorta or subclavian or axillary arteries that would prevent safe device placement, including aneurysms, significant tortuosity, or calcifications
    3. Axillary artery anatomy that would preclude safe placement of a 10F sheath including severe obstructive calcification or severe tortuosity
    4. Iliofemoral artery anatomy that would preclude safe placement of a 16F introducer sheath including severe obstructive calcification or severe tortuosity
    5. Known connective tissue disorder (e.g. Marfan Syndrome) or other aortopathy at risk of vascular injury
    6. Prior endovascular surgery or percutaneous intervention involving the thoracoabdominal aorta or a subclavian/axillary artery or history of aortic dissection
11. Severe aortic stenosis
12. Known or suspected contrast induced nephropathy
13. Absolute contraindications or allergy to iodinated contrast that cannot be adequately treated with pre-medication
14. Absolute contraindications or allergy to unfractionated heparin (e.g., heparin-induced thrombocytopenia) or device materials (e.g. nickel, titanium) that cannot be adequately treated with pre-medication
15. Known hematologic diseases such as leukemia, any coagulopathy or hypercoagulable state, sickle cell anemia or thalassemia
16. Presence of any one of the following risk factors for indications of severe end organ dysfunction or failure:

    1. Liver disease (cirrhosis of the liver [Child-Pugh class B or C]) or shock liver
    2. History of severe chronic obstructive pulmonary disease (COPD) defined by FEV1/FVC less than 0.7, and FEV1 less than 50% predicted
    3. Prior kidney transplant, isolated single kidney, stage V Chronic Kidney Disease (eGFR ≤15) at admission OR use of dialysis, continuous renal replacement therapy (CRRT) or aquapheresis (ultrafiltration) in last 90 days
17. Cardiac imaging evidence of intracardiac mass, thrombus, or vegetation
18. Symptomatic carotid or vertebral artery disease or successful treatment of carotid stenosis within 90 days prior to the index procedure
19. Active infection not controlled with antibiotic therapy
20. Suspected or known pregnancy. Women of child-bearing age should have a negative pregnancy test.
21. Body mass index (BMI) over 40 kg/m2
22. Unable or unwilling to undergo screening, device implant and retrieval procedures, and 30-day follow-up
23. Currently participating in an investigational drug or another device study that may influence the data collected for this study. Observational studies are not considered an exclusion
24. Subject has other medical, social or psychological problems that, in the opinion of the Investigator, compromises the subject ability to give written informed consent and/or to comply with study procedures
25. Active SARS-CoV-2 infection (Coronavirus-19 [COVID-19]) or previously diagnosed with COVID-19 with sequelae that could confound endpoint assessments

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Estimated)
Dates: Start 2024-08 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Device safety defined as freedom from serious in-hospital procedure or device-related adverse event (AE) | Baseline to 30-day Follow-Up
Technical success defined as successful device deployment, ability to deliver the treatment and remove the device | Baseline to 30-day Follow-Up
Assisted decongestion success defined as increase in the average hourly rate of urine output during the first 24 hours of ModulHeart-assisted decongestive therapy compared to the last 24 hours of diuretic therapy prior to pump implant | Baseline to 1 day of ModulHeart-assisted decongestive therapy

SECONDARY OUTCOMES:
Change in urine output | Baseline to end of ModulHeart therapy (up to 3 days)
Change in net fluid loss | Baseline to end of ModulHeart therapy (up to 3 days)
Change in natriuresis | Baseline to end of ModulHeart therapy (up to 3 days)
Change in creatinine clearance | Baseline to end of ModulHeart therapy (up to 3 days)
Change in N-terminal pro-B type natriuretic peptide (NT-pro BNP) | Baseline to end of ModulHeart therapy (up to 3 days)
Change in body weight | Baseline to end of ModulHeart therapy (up to 3 days)
Change in thermodilution cardiac output | Baseline to end of ModulHeart therapy (up to 3 days)
Change in right atrial pressure | Baseline to end of ModulHeart therapy (up to 3 days)
Change in mean pulmonary artery pressure | Baseline to end of ModulHeart therapy (up to 3 days)

CONTACTS AND LOCATIONS:
Locations (5):
- The Victorian Heart Hospital, Clayton, Victoria, Australia
- Georgia (4):
  - Emergency Cardiology Center by Academician G. Chapidze, Tbilisi
  - Israeli-Georgian Medical Research Clinic Helsicore, Tbilisi
  - Tbilisi Heart and Vacular Clinic, Tbilisi
  - Tbilisi Heart Center, Tbilisi

IPD SHARING:
Plan to Share IPD: No